CLINICAL TRIAL: NCT06125067
Title: Comparison of the Efficacy of Fascia Iliaca Compartment Block and IPACK Block for Postoperative Analgesia in Total Knee Arthroplasty Operation
Brief Title: Fascia Iliaca Compartment Block and IPACK Block in Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Onur Kucuk, Department of anesthesiology and reanimation, Principal Investigator, Specialist Doctor, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2012-KAEK-15/2719
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Arthropathy of Knee; Analgesia
Keywords: Total Knee Arthroplasty; iPACK Block; Fascia Iliaca Compartment Block; Postoperative Pain; Peripheral Nerve Block
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control Group (no peripheral block applied): No peripheral block was applied to this group and it was accepted as the control group. Standard multimodal analgesia and rescue analgesia according to NRS score were applied to each group
  Interventions: Procedure: no peripheral block
- Fascia Iliaca Compartment Block Group: Fascia Iliaca Compartment block was applied to this group under ultrasound guidance. Standard multimodal analgesia and rescue analgesia according to NRS score were applied to each group.
  Interventions: Procedure: Fascia Iliaca Compartment Block
- iPACK Block Group: iPACK block was applied to this group under ultrasound guidance. Standard multimodal analgesia and rescue analgesia according to NRS score were applied to each group.
  Interventions: Procedure: iPACK Block

INTERVENTIONS:
Procedure: no peripheral block — No peripheral block was applied. Standard multimodal analgesia method was applied.
  Groups: Control Group (no peripheral block applied)
Procedure: Fascia Iliaca Compartment Block — Fascia Iliaca Compartment Block is performed with the patient in a supine position. A high-frequency (6-14 MHz) linear ultrasound probe is positioned transversely to locate the femoral artery in the inguinal crease. The hyperechoic femoral nerve is usually visualized lateral to the femoral artery, between the iliopsoas and fascia iliaca. The probe is manoeuvred in a cranial and caudal direction to capture high-quality images of the femoral nerve and fascia iliaca. Identification of the triangular-shaped sartorius muscle and anterior superior iliac spine (ASIS) is achieved by lateral movement of the probe. Post-skin disinfection, the needle tip is directed just beneath the fascia iliaca. Local anaesthetic is administered following negative pressure aspiration into the area. The local anaesthetic spreads towards the femoral nerve medially and towards the iliac process laterally.
  Groups: Fascia Iliaca Compartment Block Group
Procedure: iPACK Block — During the iPACK procedure, the patient assumes a supine position with the lower extremity flexed at the knee and abducted at the hip (in frog-leg position). The ultrasound transducer is placed in the lower third of the medial thigh, and then pushed backward and downward to visualize the gap between the popliteal artery and the femoral shaft, straight above the femoral condyles. After ensuring that the needle tip is placed 2 cm beyond the lateral border of the artery, local anaesthetic solution is administrated in divided doses to infiltrate the tissue space. The needle is then withdrawn after confirming negative aspiration.
  Groups: iPACK Block Group

SUMMARY:
The investigators sought to compare the effectiveness of postoperative pain control between the standard intravenous multimodal analgesia procedure used in managing patients undergoing total knee surgery, who experience severe postoperative analgesia needs, and multimodal analgesia procedures that incorporate ultrasound-guided peripheral nerve blocks (Fascia Iliaca Compartment Block or iPACK Block) during postoperative follow-up. The aim is to determine which procedure is more effective.

DETAILED DESCRIPTION:
All patients who received a total knee replacement surgery conducted by orthopaedic surgeons at the operating theatre of Health Sciences University Ankara Atatürk Sanatorium Training and Research Hospital and underwent postoperative pain assessment by anaesthetists will be retrospectively reviewed as part of the study.

Postoperative pain management follow-up for patients who have undergone surgical procedures at Anaesthesiology and Reanimation Clinic is standard practice during patients hospitalization. Patients who have undergone painful and significant surgical procedures are typically given postoperative patient-controlled analgesia devices and are administered intravenous painkillers that are under the patient's control. As part of multimodal analgesia procedure, the investigators apply peripheral nerve blocks routinely to eligible patients, provided that the necessary criteria are met. Once the postoperative Anesthesiology and Reanimation clinic's follow-up form, the regional anaesthesia follow-up form, is completed, patients receive coordinated follow-up care from anaesthesiologists and surgical physicians in postoperative ward to monitor analgesic requirements and increase patient satisfaction. Hourly monitoring ensures that patients receive optimal care.

The aims of study to examine the effectiveness of these procedures. The investigators will include all patients who received elective total knee arthroplasty surgery in the operating room of Ankara Atatürk Sanatorium Training and Research Hospital within the past year (between 01 March 2022 and 31 March 2023) in retrospective file review and postoperative pain follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone elective total knee surgery
* ASA I-III patients

Exclusion Criteria:

* Those <30 kg
* People under 18 years of age
* Patients with missing follow-up forms
* Patients with a history of chronic opioid or corticosteroid use
* Patients with a history of inflammatory gonathrosis
* Patients with synovectomy operation history

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In our study, which is planned as a retrospective file scanning and postoperative regional anesthesia follow-up form review, all patients who have undergone elective total knee arthroplasty surgery of Ankara Atatürk Sanatorium Training and Research Hospital in the last 1 year (between 01 March 2022 and 31 March 2023) will be included in the study. It is planned to examine 120 patient files in total.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | postoperative 24 hours score change
  NRS was used to assess postoperative pain. The NRS is a segmented numerical version of the visual analog scale (VAS), in which the respondent chooses an integer (0-10 integer) that best reflects the intensity of his pain. It is considered a one-dimensional measure of pain intensity in adults. It is an 11-point numerical scale. It ranges from "0" representing no pain to "10" representing extreme pain.

SECONDARY OUTCOMES:
5-point likert satisfaction scale | postoperative 24th hour
  The patient's satisfaction with postoperative pain treatment will be recorded. 5 options; very dissatisfied, dissatisfied, neither dissatisfied or satisfied, satisfied, very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Onur KÜÇÜK, specialist, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No